CLINICAL TRIAL: NCT07082556
Title: Does Percutaneous Neuromodulation Promote Recovery in Hockey Players With Grade 0 Adductor Injuries?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Dr. Pablo Herrero Gallego, Principal Investigator, Universidad de Zaragoza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NMP-e_hockey_aductores
Record Dates: First submitted 2025-06-27; First posted 2025-07-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Grade 0 Adductor Injurie
Keywords: Neromodulation; Percutaneous; Ultrasound; Obturator nerve; hockey players

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- US-guided PNM (Experimental): Each participant will be treated with US-guided PNM targeting the anterior branch of the obturator nerve.
  Interventions: Other: US-guided PNM

INTERVENTIONS:
Other: US-guided PNM — Stimulation will be applied for 15 minutes at 4 Hz, using a 250 ms pulse duration.

SUMMARY:
Ice hockey is a widely practiced sport, particularly in North America and Europe, with over 2,500 professional players in North America and approximately 2,000 in Europe. Its global expansion has extended participation to regions such as Africa and Australia. This sport demands high physical performance, speed, strategy, and specific preparation to prevent injuries. The most common injuries include muscular and joint trauma, especially in the knees, shoulders, and groin region, where "groin pain" is a frequent issue.

Injuries to the hip joint, such as femoroacetabular impingement (FAI), acetabular labrum and cartilage lesions, and intra-articular loose bodies, are prevalent. Extra-articular injuries primarily involve the adductor and abdominal muscles. The biomechanics of ice skating require repetitive and forceful hip movements, increasing eccentric load on the adductors, particularly at higher skating speeds, thereby raising the risk of strains.

Studies have shown that the adductor muscles, particularly the adductor longus, are the most frequently injured. Risk factors include a history of previous injury, high training intensity, strength imbalances between adductors and abductors, and inadequate preseason preparation. A critical threshold is the adductor/abductor strength ratio: if it falls below 80%, the risk of injury increases 17-fold.

Invasive physiotherapy has gained prominence as an effective option for the treatment and prevention of such injuries. Ultrasound-guided invasive techniques, such as ultrasound-guided percutaneous neuromodulation (US-guided PNM), have demonstrated the ability to reduce muscle stiffness, improve intra- and intermuscular coordination, and enhance endurance. These techniques have shown greater efficacy than conventional methods, contributing to improved athletic performance and reduced injury risk.

US-guided PNM is a minimally invasive technique that delivers electrical stimulation via needles placed under ultrasound guidance near peripheral nerves or motor points. The stimulation is adjusted according to therapeutic goals, whether to reduce pain, improve neuromuscular function, or modulate muscle tone. Its efficacy has been documented in studies showing improvements in flexibility, strength, and post-exertion recovery, with effects observed even in the contralateral limb, attributed to the crossover phenomenon.

Given the high incidence of adductor injuries among hockey players and the associated risk factors, this clinical study aimed to evaluate the effectiveness of a single session of US-guided PNM in players with grade 0 (muscle contracture) injuries of the adductor muscles. Three primary variables were assessed: muscle strength (Adductor Squeeze Test), hip mobility (Bent Knee Fall Out Test), and subjective pain (VAS scale), both in daily activities and during on- and off-ice training.

DETAILED DESCRIPTION:
Ice hockey is one of the most widely followed and practiced professional sports in both North America and Europe, with a high number of registered players in both regions. The sport continues to expand globally, reaching nations in diverse parts of the world such as Africa and Australia. In North America, the National Hockey League (NHL) is the top professional league, comprising 32 teams and approximately 750 active players, supported by minor leagues like the American Hockey League (AHL) and the East Coast Hockey League (ECHL), which together include over 1,800 players. Consequently, the total number of professional players in North America exceeds 2,500 athletes. The number of adult professional and non-professional registered players in North America is approximately 230,000 (IIHF Survey). In Europe, ice hockey is structured into various top-level national championships, which collectively account for 1,500 to 2,000 professional players. The total number of adult registered players in this region is approximately 83,000. Therefore, it is estimated that the number of professional ice hockey players worldwide is around 4,000 to 4,500, confirming the strong presence and ongoing development of the sport at an international scale.

This sport requires the integration of several key elements, including physical intensity, speed, and strategy, demanding a high level of athletic preparation and close attention to injury prevention. A professional player must train specifically to develop explosive power, static and dynamic balance, and anaerobic endurance in order to accelerate rapidly, change direction with agility, and maintain puck control under pressure. Constant physical contact and the risk of high-speed collisions increase the likelihood of injuries, with frequent muscular and joint trauma, particularly in the knees and shoulders, as well as concussions caused by impacts with boards or other players. In their systematic review, Bérubé et al. aimed to determine the most common orthopedic injuries among NHL players. The most studied anatomical regions were the hip and pelvis (24%), followed by the ankle (10%), knee (10%), shoulder (7%), and foot (7%).

This sport imposes intense physical demands that generate specific biomechanical requirements, particularly on the lower limbs, often forcing the hip to perform repetitive movements beyond its physiological limits. Players are frequently affected by groin injuries or hip joint pain, which may prevent them from competing. So-called "groin pain" is a widespread issue among ice hockey players and may have an acute or chronic etiology, originating from extra-articular or intra-articular structures that produce varying symptoms. Kuhn et al. identified the most common intra-articular injuries as acetabular labrum tears, femoroacetabular impingement (FAI) - both "cam" and "pincer" types - cartilage degeneration, and intra-articular loose bodies. Among these, acetabular labrum tears had the highest incidence (69.1%), followed by cartilage injuries (13.8%), loose bodies (6.3%), and FAI (5.3%). The most frequent extra-articular conditions include adductor muscle and abdominal injuries.

Hip adduction is performed by six muscles: adductor longus, adductor magnus, adductor brevis, gracilis, obturator externus, and pectineus. All are innervated by the obturator nerve (both anterior and posterior branches), except for the adductor magnus, which also receives innervation from the sciatic nerve, and the pectineus, which also receives fibers from the femoral nerve.

From a biomechanical standpoint, skating is a biphasic movement involving single and double support phases and a swing phase. Propulsion is achieved through hip extension, abduction, and external rotation, along with knee extension. During this phase, the hip must move in flexion-extension (sagittal plane), abduction-adduction (frontal plane), and internal-external rotation (transverse plane). The adductor muscles play a key role in eccentric deceleration in the final stage of propulsion, preceding their concentric activation during leg recovery. As skating speed increases, both stride frequency and length increase, along with greater lateral hip displacement and range of motion in multiple directions. The resulting increase in hip abduction leads to greater eccentric loading on the adductors. Repeated eccentric contractions, necessary to control leg deceleration, can contribute to muscle injuries, highlighting the need for preventive strategies.

Stephen J. Nicholas reports that approximately 10% of all injuries in ice hockey involve the adductor muscle group, with a particularly high incidence among elite players. The most frequently injured muscle is the adductor longus, likely due to its superficial position, length, and mechanical disadvantage. In a study of elite Finnish players over three seasons, 43% of all muscle injuries were adductor strains. In the NHL, the incidence is 3.2 muscle injuries per 1,000 game exposures, with cases increasing in the pre-season. Serner et al. note that in sports involving rapid directional changes, adductor injuries account for most acute groin injuries, with the adductor longus involved in 87% of cases, followed by the adductor brevis (25%), pectineus (24%), and other muscles less frequently.

Key risk factors for adductor injuries include a history of prior injuries and high levels of competition, where training intensity and volume place greater strain on the adductors. Absolute and relative adductor strength, particularly the adductor-to-abductor strength ratio, is critical. Muscle imbalances caused by adductor weakness significantly increase the likelihood of strain injuries. These assumptions are supported by Tyler et al., who found that previous injuries increase the risk of recurrence by 2.4 times. The higher the competition level, the greater the training intensity and volume to which the adductors are subjected, and consequently, the higher the injury risk. Injured athletes show an average of 18% less adductor strength compared to non-injured athletes, and the adductor/abductor strength ratio is reduced (78% vs. 95%). When this ratio drops below 80%, the injury risk increases 17-fold. Additionally, inadequate sport-specific training, particularly during the pre-season, may predispose athletes to injury due to insufficient muscular preparation.

Advancements in invasive physiotherapy techniques have opened new possibilities for treatment and recovery optimization, significantly impacting both rehabilitation and injury prevention in sports. Owing to their targeted, precise, effective, and safe mechanisms of action, some of these techniques have become valuable tools to enhance athletic performance, reduce injury risk and recurrence, and improve the management of musculoskeletal conditions.

Studies on muscle flexibility have confirmed that ultrasound-guided invasive techniques significantly reduce muscle stiffness with immediate effects. Additional benefits include improvements in intra- and intermuscular coordination and muscle endurance, which more effectively reduce fatigue and enhance stability compared to stretching and eccentric exercises. Compared to other physiotherapy approaches, invasive techniques have shown superior results, making them a promising option in both rehabilitation and prevention. These effects help maintain muscular balance, preventing overload and compensatory patterns.

In this context, ultrasound-guided percutaneous neuromodulation (US-guided PNM) may be considered an innovative and promising approach to improve athletes' health and performance. Although the quantity and quality of scientific evidence are still limited, further studies are necessary to validate current findings and better define the clinical applications of these techniques.

US-guided PNM is a minimally invasive technique involving electrical stimulation applied via fine needles inserted under ultrasound guidance near peripheral nerves or motor points. The procedure begins with ultrasound localization of the target area, followed by needle insertion at an optimal angle and direction for safe access. A surface electrode is then placed to complete the circuit and allow the generation of a biphasic electrical field. Electrical stimulation is applied with adjustable parameters, typically at low frequencies (2-10 Hz) for muscle relaxation or high frequencies (50-100 Hz) for pain control. The stimulation duration ranges from 15 to 30 minutes, depending on therapeutic objectives. The benefits of this technique include pain reduction, improved neuromuscular function, and muscle tone modulation. As such, US-guided PNM can be considered effective in managing musculoskeletal and neurological conditions.

In their systematic review, Fidalgo et al. highlight the effects of US-guided PNM, including enhanced muscle contraction, increased motor unit recruitment, and improved isometric strength - all valuable for athletes and individuals with muscular weakness. Additionally, US-guided PNM can improve muscle flexibility by reducing stiffness and increasing range of motion, especially in the hip and knee. It also helps decrease muscle fatigue, optimize post-exertion recovery, and enhance neuromuscular efficiency.

De-La-Cruz-Torres et al. demonstrated that US-guided PNM significantly improves hamstring flexibility, suggesting a central neuromodulatory effect. These changes may reduce the risk of injury, supporting its use in athletes and/or patients with motor limitations. The study also found improvements in the contralateral limb, explained by the "crossover" effect. According to the authors, stimulation of one limb may induce adaptations in the opposite limb via activation of central and peripheral neuromodulatory pathways.

Considering the high incidence of adductor muscle injuries among elite ice hockey players and the predictive risk factors related to isolated and combined agonist-antagonist strength ratios, the aim of this clinical study was to evaluate the effectiveness of a single US-guided PNM treatment on functional recovery in players with grade 0 (muscle contracture) injuries of the adductor muscles.

The specific objectives were as follows:

To analyze changes in adductor muscle strength following a single US-guided PNM session.

To evaluate changes in hip joint mobility after a single US-guided PNM session.

To determine the effect of US-guided PNM on pain perception in various contexts: daily life activities, on-ice training, and off-ice training, after a single intervention.

The variables analyzed in this study include: mean subjective pain measured using the Visual Analogue Scale (VAS), hip mobility assessed with the Bent Knee Fall Out Test (BKFO) and measured in centimeters, and adductor muscle strength evaluated with the Adductor Squeeze Test (AST), expressed in kilograms.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Pain in the adductor region
* Clinical diagnosis with ultrasound confirmation of the absence of structural damage, consistent with a grade 0 muscle injury (contracture) localized in the adductors

Exclusion Criteria:

* Presence of muscle injuries above grade 0
* Concomitant neurological, systemic, or orthopedic conditions
* Recent application of neuromodulation techniques or other similar treatments performed by healthcare professionals within the last 7 days
* Belonephobia (fear of needles)
* Infections or skin disorders localized in the inguinal region

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2025-06-27 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
VAS (ADL) | 2 times, immediately pre-intervention and immediately after the first training posterior to the intervention.
  Pain during the activities of the daily life. This variable will be assessed through the Visual Analogue Scale (0-10 points)
VAS (ON ice) | 2 times, immediately pre-intervention and immediately after the first training posterior to the intervention.
  Pain during hockey training on ice. This variable will be assessed through the Visual Analogue Scale (0-10 points)
VAS (OFF ice) | 2 times, immediately pre-intervention and immediately after the first training posterior to the intervention.
  Pain during training out of the ice. This variable will be assessed through the Visual Analogue Scale (0-10 points)

SECONDARY OUTCOMES:
Maximum Isometric Strength. Hip Adductors | 2 times, immediately pre-intervention and immediately post-intervention
  This variable will be assessed using the "Adductor Squeeze Test" and a dynamometer (K-Force Push).
Passive hip mobility | 2 times, immediately pre-intervention and immediately post-intervention.
  Passive hip mobility in flexion, abduction, and external rotation: this variable will be assessed using the Bent Knee Fall Out Test (BKFO).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Herrero, Physiotherapist, Study Director — Universidad de Zaragoza
Locations (1):
- University of Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a reasonable request contacting with the main author once data has been published.
  Anyway, Individual participant data (IPD) will be shared with other researchers in accordance with data sharing protocols and participant consent, ensuring confidentiality and ethical considerations are maintained.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once research has been published
Access Criteria: Study protocol will be publish in a scientific journal